CLINICAL TRIAL: NCT05911464
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10386 in Participants With Advanced Solid Tumors
Brief Title: A Phase I Study of HS-10386 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10386-101
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumors; Immuno-Oncology Therapy; Immunotherapy; Immune Checkpoint Inhibitor; PD-1; PD-L1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10386 (Experimental): Participants will receive HS-10386 once daily. The duration of each treatment cycle is 21 days.
  Interventions: Drug: HS-10386

INTERVENTIONS:
Drug: HS-10386 — Starting dose 10 mg, administered once daily. If tolerated, subsequent cohorts will test increasing doses of HS-10386, until a maximum tolerated dose (MTD) or maximum applicable dose (MAD) is defined

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, and preliminary anti-tumor activity of HS-10386 in participants with advanced solid tumors who have failed prior treatments.

DETAILED DESCRIPTION:
This is a phase I open label, multicenter clinical study to evaluate the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of HS-10386 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years old.
2. Histologically or cytologically documented, incurable or metastatic solid tumors for which standard treatment either does not exist or has proven ineffective or unavailable or intolerable.
3. At least one measurable lesion per RECIST v1.1.
4. Willingness to provide fresh or archival tumor biopsy sample.
5. An Eastern Cooperative Oncology Group (ECOG) performance status equal to 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
6. Willingness to use adequate contraceptive measures throughout the study.
7. Ability to comprehend and willingness to sign a written ICF for the study.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with systemic immunotherapy.
   2. Treatment with anticancer medications or investigational drugs within protocol-defined intervals prior to the first scheduled dose of HS-10386.
2. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 except for alopecia.
3. Known additional malignancy.
4. History or risk of autoimmune disease.
5. Known primary CNS malignancy or symptomatic CNS metastases. Patients with asymptomatic CNS metastases may be enrolled after consultation.
6. Inadequate bone marrow reserve or organ function.
7. Clinically significant cardiac disease.
8. Any evidence of severe or uncontrolled systemic diseases
9. Severe infections within 4 weeks prior to the first scheduled dose or symptoms of infection within 2 weeks prior to prior to the first scheduled dose.
10. History of organ transplantation or any medical condition requiring the use of systemic immunosuppressive medications.
11. Active HBV or HCV infection that requires treatment.
12. Known history of HIV.
13. Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
14. Administration of a live, attenuated vaccine within 4 weeks prior to the first scheduled dose or anticipation that such a live attenuated vaccine will be required during the study.
15. History of severe anaphylaxis or allergic to any of the components of HS-10386.
16. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) or Maximum Applicable Dose (MAD) (Dose Escalation Phase) | Up to 21 days from the first dose
  MTD is defined as the dose level immediately below that at which 2 or more patients exhibit dose limiting toxicity. MAD is defined as the maximum administered dose, when MTD is not reached.
Objective Response Rate (ORR) defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (Dose Expansion Phase) | Every 6 weeks for the duration of study participation; estimated to be 12 months.
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | From Informed consent until the end of the follow-up period which is defined as 28 days (+7 days) after study treatment is discontinued.
  The number and percentage of patients that experience an AE. The severity of AEs are assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Cmax of HS-10386 | Approximately 1 month.
  Cmax is defined as the maximum observed plasma or serum concentration.
Tmax of HS-10386 | Approximately 1 month.
  Tmax is defined as the time to maximum concentration.
λz of HS-10386 | Approximately 1 month.
  λz is defined as the apparent terminal-phase disposition rate constant.
t1/2 of HS-10386 | Approximately 1 month.
  t1/2 is defined as the apparent terminal-phase disposition half-life.
AUC0-t of HS-10386 | Approximately 1 month
  AUC0-t is defined as the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
CL/F of HS-10386 | Approximately 1 month.
  CL/F is defined as the apparent oral dose clearance.
ORR defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (Dose Escalation Phase) | Every 6 weeks for the duration of study participation; estimated to be 12 months.
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression.
Disease Control Rate (DCR) | Every 6 weeks for the duration of study participation; estimated to be 12 months.
  The DCR is defined as the percentage of patients with a best overall response of CR, PR, or SD.
Duration of Response (DoR) | Every 6 weeks for the duration of study participation; estimated to be 12 months.
  DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Progression-Free Survival (PFS) | Every 6 weeks for the duration of study participation; estimated to be 12 months.
  PFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to PD or death from any cause.
Overall Survival (OS) (Dose Expansion Phase) | From the time of randomization to death due to any cause, approximately 3 years.
  OS is deﬁned as the time from randomization to death due to any cause.
The correlation between PD-L1 expression and efficacy of HS-10386 | Approximately 3 years.
  The study will collect tumor tissue samples during screening period and after the treatment. Stratified analysis of the efficacy endpoint of HS-10386 (such as object response, DoR, PFS, etc.) by PD-L1 expression level will be performed to assess the correlation between PD-L1 expression as biomarker and study dose and effeicacy of HS-10386.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Dr., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China